CLINICAL TRIAL: NCT06644664
Title: The Effect of Nicotine and Tobacco Message Framing on Use Among Diverse Groups of Young Adults: Aim 3 Randomized Control Trial (RCT)
Brief Title: Nicotine and Tobacco Message Framing to Change Smoking Behavior in Diverse Groups of Young Adult Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joanne Patterson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-23436; NCI-2024-04955 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R00CA260718 (NIH)
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Tobacco-Related Carcinoma
Keywords: Sexual and Gender Minorities; Health Communication; Tobacco Products; Cigarettes; Electronic Nicotine Delivery Systems; E-cigarettes; young adult; text messaging
MeSH Terms: conditions — Coitus; Vaping | interventions — Interviews as Topic; Smoking Devices

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blinded to their randomization category (absolute risks, relative risks, or control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (Absolute Risk messages) (Experimental): Participants receive AR anti-polytobacco MMS messages TIW and a check-in text message QW for a total of 6 weeks. Participants also receive smoking cessation resources via email during follow up.
  Interventions: Other: Interview; Behavioral: Smoking Cessation Intervention; Other: Survey Administration; Other: Text Message-Based Navigation Intervention
- Arm II (Relative Risk messages) (Experimental): Participants receive RR anti-polytobacco MMS messages TIW and a check-in text message QW for a total of 6 weeks. Participants also receive smoking cessation resources via email during follow up.
  Interventions: Other: Interview; Behavioral: Smoking Cessation Intervention; Other: Survey Administration; Other: Text Message-Based Navigation Intervention
- Arm III (control messages) (Active Comparator): Participants receive control MMS messages on health risks of UV/sun exposure TIW and a check-in text message QW for a total of 6 weeks. Participants also receive smoking cessation resources via email during follow up.
  Interventions: Behavioral: Health Education; Behavioral: Smoking Cessation Intervention; Other: Survey Administration; Other: Text Message-Based Navigation Intervention

INTERVENTIONS:
Behavioral: Health Education — Receive control MMS messages
  Arms: Arm III (control messages)
Other: Interview — Ancillary studies
  Arms: Arm I (Absolute Risk messages); Arm II (Relative Risk messages)
Behavioral: Smoking Cessation Intervention — Receive AR MMS messages
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Arm I (Absolute Risk messages)
Behavioral: Smoking Cessation Intervention — Receive RR MMS messages
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Arm II (Relative Risk messages)
Behavioral: Smoking Cessation Intervention — Receive smoking cessation resources
  Other Names: Smoking and Tobacco Use Cessation Interventions
Other: Survey Administration — Ancillary studies
Other: Text Message-Based Navigation Intervention — Receive check-in text message
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation

SUMMARY:
This clinical trial evaluates the effect of message framing on smoking behaviors among lesbian, gay, bisexual, transgender, queer (LGBTQ+) young adults who use nicotine and/or tobacco. Tobacco regulation has contributed to a steady decline in tobacco products designed to be smoked (combustible), but there has been an increase in the use of new tobacco products, such as electronic nicotine delivery systems (ENDS). The use of more than one tobacco product (polytobacco) is high in LGBTQ+ populations. Both LGBTQ+ people and people who engage in polytobacco use are less likely to view tobacco as harmful, which may reinforce tobacco use. Message framing includes culturally targeted messages to communicate the absolute risks (AR) and relative risks (RR) of polytobacco use. Using message framing may increase quit rates or change smoking behaviors in LGBTQ+ young adults who use nicotine and/or tobacco products.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility of delivering mobile multimedia messaging (MMS) anti-tobacco messages developed in the K99 to LGBT young adults via texting.

II. Estimate effect sizes of exposure to anti-tobacco messages on risk perceptions and tobacco use over time.

OUTLINE: Participants are randomized to 1 of 3 arms.

ARM I: Participants receive AR anti-polytobacco MMS messages 3 times a week (TIW) and a check-in text message once a week (QW) for a total of 6 weeks.

ARM II: Participants receive RR anti-polytobacco MMS messages TIW and a check-in text message QW for a total of 6 weeks.

ARM III: Participants receive control MMS messages on health risks of ultraviolet (UV)/sun exposure TIW and a check-in text message QW for a total of 6 weeks.

All participants also receive smoking cessation resources via email during follow up.

After completion of study intervention, participants are followed up at 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Self-identify as LGBTQ+
* Able to speak English fluently
* An ever user of ENDS and combustible tobacco who currently use ENDS, combustible cigarettes, or both ENDS and combustible cigarettes
* Currently reside in the United States (US)
* Have a mobile phone through a U.S. carrier with MMS messaging and can send and receive text messages for study participation
* Access to the internet with Zoom capabilities

Exclusion Criteria:

* Have a landline or Voice Over Internet Protocol (VOIP) phone number

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total tobacco cessation | At 12 weeks post-baseline
  2 items. Asks for current use of nicotine vapes and combustible cigarettes Every day, Some days, or Not at all.
Acceptability of multimedia messaging service (MMS) anti-polytobacco messages | At 6-week post-enrollment
  In a qualitative interview, Participants will be asked the following question: How did you find participating in a study with images sent via text message? How smoothly would you say it went?
Feasibility of MMS anti-polytobacco messages | At 6-weeks post-enrollment
  6 items per study arm. Experimental arms 1 and 2: 6 Yes/No questions (1 per week) checking for engagement with the study content, specifically regarding nicotine and tobacco use. Control Group: 6 Yes/No questions (1 per week) checking for engagement with the study content, specifically regarding sun safety.

SECONDARY OUTCOMES:
Switching to exclusive electronic nicotine delivery system (ENDS) use | At 6- and 12-weeks post-baseline
  2 items. Asks for current use of nicotine vapes and combustible cigarettes Every day, Some days, or Not at all.
Risk perceptions | At 6- and 12-weeks post-baseline
  3 items. 2 items on a 5 point likert scale where 1= Not at all harmful and 5= Extremely harmful. How harmful do you think nicotine vapes, e-cigarettes, or other electronic products are to health? How harmful do you think cigarettes are to health?; 1 item with 3 response options: Less harmful, About the same, More harmful. Is using nicotine vapes, e-cigarettes or other electronic nicotine products less harmful, about the same, or more harmful than smoking cigarettes?
Behavioral intentions | Difference between conditions in behavioral intentions from screener, and at 6 and 12-week post baseline
  2 Items. Are you seriously thinking of quitting nicotine vapes? and Are you seriously thinking of quitting cigarettes? 5 response options: Yes, within the next 30 days; Yes, within the next 6 months; Yes, within the next year; Yes, but not within the next year; No, not thinking of quitting.
Serious quit attempts | Difference between conditions in quit attempts from screener, and at 6 and 12-week post baseline
  2 items. During the PAST 12 MONTHS, how many times have you stopped vaping nicotine for 1 day or longer because you were trying to quit? and During the PAST 12 MONTHS, how many times have you stopped vaping nicotine for 1 day or longer because you were trying to quit? 5 response options: None; 1-2 times; 3-5 times; 6-10 times; More than 10 times

CONTACTS AND LOCATIONS:
Overall Officials: Joanne G Patterson, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Our Health Matters — https://u.osu.edu/lgbtqhealthequity/research/my-health-matters/